CLINICAL TRIAL: NCT05665907
Title: Evaluation of Executive Functions in Children With Cochleovestibular Deficit
Acronym: Vestibulex
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220224; IDRCB: 2022-A00160-43 (Registry Identifier: French Health Authority)
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-11

CONDITIONS: Vestibular Function; Hearing Loss; Cognitive Function; Executive Function
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with vestibular dysfunction with hearing loss: children with vestibular dysfunction with hearing loss
  Interventions: Other: Questionnaire BRIEF (Behavioral Rating Inventory of Executive Function)
- children with vestibular dysfunction with normal inner ear function: children with vestibular dysfunction with normal inner ear function
  Interventions: Other: Questionnaire BRIEF (Behavioral Rating Inventory of Executive Function)

INTERVENTIONS:
Other: Questionnaire BRIEF (Behavioral Rating Inventory of Executive Function) — Questionnaire BRIEF (Behavioral Rating Inventory of Executive Function)

SUMMARY:
Vestibular system activity supports many functions ranging from gaze stabilization and postural control to high-level cortical functions involving spatial cognition, body perception, verticality perception, orientation, navigation, and spatial memory. Few studies have assessed the impact of a vestibular deficit on executive functions taking into account the simultaneous existence of sensorineural deafness in a child population. The BRIEF questionnaire (Behavioral Rating Inventory of Executive Function) allows a parental assessment of executive functions and is validated from the age of 5. Children were recruited from a pediatric population followed in the Ear Nose and Throat (ENT) department for audio-vestibular assessment and BRIEF questionnaire was completed by the accompanying parent.

DETAILED DESCRIPTION:
Vestibular system activity supports many functions ranging from gaze stabilization and postural control to high-level cortical functions involving spatial cognition, body perception, verticality perception, orientation, navigation, and spatial memory. Few studies have assessed the impact of a vestibular deficit on executive functions taking into account the simultaneous existence of sensorineural deafness in a child population. The BRIEF questionnaire (Behavioral Rating Inventory of Executive Function) allows a parental assessment of executive functions and is validated from the age of 5. Children were recruited from a pediatric population followed in the Ear Nose and Throat (ENT) department for audio-vestibular assessment and BRIEF questionnaire was completed by the accompanying parent.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 5 years < 18 years with vestibulopathy confirmed during an ENT consultation
* Affiliated to the social security system
* Holders of parental authority and Patients informed and not opposed to participating in the research
* Mastery of the French language by patients and their parents

Exclusion Criteria:

* Refusal to participate
* Existence of another neurodevelopmental pathology or specific cognitive disorder

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children with vestibular dysfunction, with hearing loss or normal inner ear function
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Global scores on the BRIEF (Behavioral Rating Inventory of Executive Function) questionnaire | 1 year
  Comparison of global scores obtained in children with vestibular dysfunction, with hearing loss or normal inner ear function

CONTACTS AND LOCATIONS:
Overall Officials: Audrey MAUDOUX, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided